CLINICAL TRIAL: NCT02134314
Title: Assessing Safety and Efficacy of Preoperative and Post-Transplant C1 Inhibitor (Berinert®) vs. Placebo in Recipients of a Renal Allograft From Deceased High Risk Donors and Its Impact on DGF and IRI
Brief Title: C1INH Inhibitor Preoperative and Post Kidney Transplant to Prevent DGF & IRI
Acronym: C1INHDGF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Stanley Jordan, MD, Medical Director, Kidney Transplant Program; Director of Transplant Immunology and Nephrology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C1INH (Berinert) for DGF; IND15806 (Other: FDA)
Record Dates: First submitted 2014-02-19; First posted 2014-05-09 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: End Stage Renal Disease; Kidney Failure; Delayed Graft Function; Ischemic Reperfusion Injury
Keywords: ESRD (End Stage Renal Disease); CKD (Chronic Kidney Disease); Kidney Transplant; ECD; delayed graft function; chronic kidney disease; expanded-criteria donor; end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Delayed Graft Function; Renal Insufficiency, Chronic | interventions — Complement C1 Inhibitor Protein; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C1-Inhibitor (Berinert) (Human) (C1INH) (Experimental): 35 patients will receive C1 esterase inhibitor in addition to standard of care immunosuppressive therapy.
  Interventions: Drug: C1 Esterase Inhibitor
- Normal Saline (Placebo Comparator): 35 patients will receive placebo in addition to standard of care immunosuppressive therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C1 Esterase Inhibitor — C1 Esterase Inhibitor 50 units per kilogram intravenous infusion administered on day of transplant, and another dose at 24 hours post-operatively. Total: 2 doses
  Other Names: Berinert (C1INH)
  Arms: C1-Inhibitor (Berinert) (Human) (C1INH)
Drug: Placebo — Placebo medication identical to study drug (C1 esterase inhibitor) volume will be administered on day of transplant, and another dose at 24 hours post-operatively. Total: 2 doses
  Other Names: Normal Saline (0.9%NaCl)
  Arms: Normal Saline

SUMMARY:
The use of C1INH (Berinert) in patients receiving deceased donor kidney transplants with high risk for delayed graft function (DGF) may show significant improvement in outcomes post transplant compared with patients that do not receive C1INH treatment. Complement activation has been detected in animal models and human kidneys with ischemic reperfusion injury (IRI) and inflammatory cell infiltrates. By blocking complement activation the investigators hope to improve kidney graft function post transplant in these recipients.

DETAILED DESCRIPTION:
Early graft function has a long-term effect on graft survival. Poor early graft function and delayed graft function (DGF) contributes to decreased short- and long-term patient and graft survival, increased incidence of acute rejection, prolonged hospitalization, and higher costs of transplantation. Although multiple factors contribute to the impaired graft function, ischemia-reperfusion injury (IRI) is the underlying pathophysiology leading to poor early graft function and DGF. A >35% incidence of DGF has remained constant over time despite significant improvements in immunosuppressive strategies and patient management. This may be due to increased use of kidneys from "extended-criteria" and/or non-heart-beating donors, where even greater rates (>60%) of DGF have been reported.

More than 96,680 people are currently waiting for a kidney transplant in the United States (United Network for Organ Sharing (UNOS); UNOS.org 3/22/13). Of the 15,092 kidney transplants performed in the US in 2011, ~11,000 (62%) were from deceased donors. Of these, approximately 17% were from expanded-criteria donors. The USRDS reports that more than 50% of patients on the waiting list are willing to accept a kidney from an expanded-criteria donor (ECD) or donors after cardiac death (DCD).

From the investigators previous studies with C1INH (Berinert®) for prevention of antibody mediated rejection (ABMR), the investigators noted that no patients developed ABMR during treatment with C1INH, the investigators also noted a near significant reduction in DGF due to IRI (ClinicalTrials.gov(NCT01134510), FDA Investigational New Drug (IND#): 14363). These findings suggest an important role for complement in the mediation of IRI and that inhibition of early complement activation using C1INH in patients receiving at risk kidneys for IRI should reduce this costly and often devastating complication of kidney transplantation. In addition, numerous other studies in animal models have shown dramatic improvements in IRI models with the use of C1INH. Complement activation is detectable in animal and in human kidneys models after IRI and experimental data suggests that use of C1INH prior to induction of IRI significantly reduces IRI as well as inflammatory cell infiltrates. Based on this, the investigators hypothesize that the use of C1INH in patients receiving deceased donor (DD) kidney transplants with high risk for DGF will show significant reductions in DGF and improved outcomes post-transplant compared with patients receiving DD transplants who do not receive C1INH treatment. Here, the investigators propose to investigate the application of pre-operative and post-transplant doses of C1INH (Berinert®) vs. placebo in adult subjects receiving a DD renal allograft considered at high-risk for IRI and DGF. The investigators hypothesize that C1INH treated patients will demonstrate improved function of the kidney allograft compared to placebo, with equivalence in safety. The primary objectives of this study are: Using a double blinded, placebo controlled format, the investigators will:

1. Evaluate and compare the safety of C1INH (50 units/kilogram, round to the nearest 500 unit) administered pre-transplant and 24 hrs post-transplant in recipients of kidney allografts from high risk for IRI deceased donors.

The secondary objectives are to:

1. On the basis of safety and efficacy, determine appropriate Berinert® study dose for Phase III investigation, and
2. Determine appropriate endpoint choice for Phase III investigation.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 yrs of age; recipient of ECD/DCD/ECD&DCD with risk index 3-8 for DGF based on specific criteria
* recipient who are ABO compatible with donor allograft
* pretransplant with meningococcal vaccination
* understand and sign a written consent prior to any study specific procedure.

Risk index (minimum 3- maximum 8):

DGF scale: Donor Age (<40yr = 0, 41-49yr = 1, 50-54yr = 2, 55-59yr = 3, >60yr=6), Cold Ischemia Time (0-12= 0, 13-18=1, 19-24=2, 24-30=3, 31-36=4, >37=6; Recipient Race (nonblack = 0, black =1); Donor death due to Cerebrovascular Accident (CVA) (donor age <50yrs = 0, donor age >50yrs = 3).

Exclusion Criteria:

* patients with known prothrombotic disorder (e.g. factor V leiden)
* history of thrombosis or hypercoagulable state excluding access clotting
* history of administration of C1INH containing products or recombinant C1INH within 15 days prior to study entry
* patients with known contraindication to treatment with C1INH
* patients with abnormal coagulation function (INR >2, partial thromboplastin time (PTT) > 50, platelets <80,000)
* who are not on anti-coagulation
* patients with known active presence of malignancies
* Polymerase chain reaction (PCR) positive for hep B/hep C/or HIV
* preemptive kidney transplantation recipient
* recipients of multi-organ transplants (kidney and any other organ)
* recipients of kidney allograft from DD who: cold ischemia time (CIT) <18h, terminal serum creatinine </= 1mg/dl, recipient of kidney allograft that was on pump preservation for any period prior to transplantation, recipient of kidney allograft from a living donor, female subject who are pregnant or lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09; Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley C Jordan, MD, Principal Investigator — Cedars-Sinai Medical Center, Los Angeles, CA; Ashley Vo, PharmD, Study Director — Cedars-Sinai Medical Center, Los Angeles, CA
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Dalle Lucca JJ, Li Y, Simovic M, Pusateri AE, Falabella M, Dubick MA, Tsokos GC. Effects of C1 inhibitor on tissue damage in a porcine model of controlled hemorrhage. Shock. 2012 Jul;38(1):82-91. doi: 10.1097/SHK.0b013e31825a3522. PMID 22683724
- [Background] Pascual J, Zamora J, Pirsch JD. A systematic review of kidney transplantation from expanded criteria donors. Am J Kidney Dis. 2008 Sep;52(3):553-86. doi: 10.1053/j.ajkd.2008.06.005. PMID 18725015
- [Background] Castellano G, Melchiorre R, Loverre A, Ditonno P, Montinaro V, Rossini M, Divella C, Battaglia M, Lucarelli G, Annunziata G, Palazzo S, Selvaggi FP, Staffieri F, Crovace A, Daha MR, Mannesse M, van Wetering S, Paolo Schena F, Grandaliano G. Therapeutic targeting of classical and lectin pathways of complement protects from ischemia-reperfusion-induced renal damage. Am J Pathol. 2010 Apr;176(4):1648-59. doi: 10.2353/ajpath.2010.090276. Epub 2010 Feb 11. PMID 20150432
- [Background] Giral-Classe M, Hourmant M, Cantarovich D, Dantal J, Blancho G, Daguin P, Ancelet D, Soulillou JP. Delayed graft function of more than six days strongly decreases long-term survival of transplanted kidneys. Kidney Int. 1998 Sep;54(3):972-8. doi: 10.1046/j.1523-1755.1998.00071.x. PMID 9734625
- See also: Cedars Sinai Medical Center Kidney Transplantation — http://cedars-sinai.edu/Patients/Quality-Measures/Clinical-Areas/Transplantation/Kidney-Transplantation.aspx
- See also: Information of C1INH (Berinert) — http://www.berinert.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- C1-Inhibitor (Berinert) (Human) (C1INH): 35 patients will receive C1 esterase inhibitor in addition to standard of care immunosuppressive therapy.
  C1 Esterase Inhibitor: C1 Esterase Inhibitor 50 units/kg intravenous infusion administered on day of transplant, and another dose 24 hours post op. Total: 2 doses
- Normal Saline: 35 patients will receive placebo in addition to standard of care immunosuppressive therapy.
  Placebo: Placebo medication identical to study drug (C1 esterase inhibitor) volume will be administered on day of transplant, and another dose 24 hours post op. Total: 2 doses
Period: Overall Study
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Started | 35 | 35
Completed | 34 | 34
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.66 (7.74) | 58.14 (11.18) | 57.9 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 20 | 22 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Patients were categorized as either African American or not African American.
  Participants
    African-American | 4 | 4 | 8
    Not African-American | 31 | 31 | 62
Diabetes [Count of Participants; unit: Participants] | 21 | 20 | 41
Donor Age [Mean (Standard Deviation); unit: years] | 49.17 (12.35) | 45.57 (15.69) | 47.37 (14.13)
Donor Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.78 (1.44) | 1.75 (1.92) | 1.77 (1.69)
Donor DCD Cause of Death [Count of Participants; unit: Participants] — The kidney transplant donor was a Donor after Cardiac Death (DCD).
  Participants | 11 | 12 | 23
Donor KDPI [Mean (Standard Deviation); unit: %] — Mean kidney transplant donor Kidney Donor Profile Index (KDPI), shown as a percentage. Kidneys with a high KDPI are associated with higher rates of DGF and worse long term survival in comparison to those with a low KDPI. In this study, the eligibility criteria included recipients of kidney allografts from ECD (or KDPI >/= 85) donors. A KDPI >/= 85 confers the highest risk for DGF and allograft loss.
  % | 67.71 (21.83) | 64.63 (25.39) | 66.17 (23.56)
Donor KDPI equal to or greater than 85% [Count of Participants; unit: Participants] — The donor's Kidney Donor Profile Index (KDPI) was equal to or greater than 85%. Mean kidney transplant donor Kidney Donor Profile Index (KDPI), shown as a percentage. Kidneys with a high KDPI are associated with higher rates of DGF and worse long term survival in comparison to those with a low KDPI. In this study, the eligibility criteria included recipients of kidney allografts from ECD (or KDPI >/= 85) donors. A KDPI >/= 85 confers the highest risk for DGF and allograft loss.
  Participants | 10 | 11 | 21
Transplant Cold Ischemia Time [Mean (Standard Deviation); unit: hours] | 18.27 (4.89) | 19.84 (6.10) | 19.06 (5.54)
Anti-HLA DSA [Count of Participants; unit: Participants] — Anti-Human leukocyte antigen (HLA) Donor Specific Antibody (DSA)
  Participants | 3 | 2 | 5
HLA Class I Antibodies Present [Count of Participants; unit: Participants] — Human leukocyte antigen (HLA) Class I Antibodies
  Participants | 2 | 1 | 3
HLA Class II Antibodies Present [Count of Participants; unit: Participants] — Human leukocyte antigen (HLA) Class II Antibodies
  Participants | 1 | 1 | 2
Treatment with Thymoglobulin at transplantation [Count of Participants; unit: Participants] — Patients who received thymoglobulin as an induction agent at transplant
  Participants | 25 | 28 | 53
Treatment with Alemtuzumab at transplantation [Count of Participants; unit: Participants] — Patients who received alemtuzumab (Campath) as an induction agent at transplant
  Participants | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Enrolled With Serum Creatinine >3mg/dL on Postoperative Day 5.
Description: Number of participants in the C1INH and placebo groups with serum creatinine >3mg/dL on postoperative day 5
Time Frame: First 7 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 34 | 35
Participants | 29 | 32

2. Primary Outcome: Number of Patients Enrolled Who Require at Least One Session of Dialysis in the First 7 Days Post Transplant.
Description: The proportion of patients enrolled who require at least one session of dialysis in the first 7 days post transplant (excluding those who are dialyzed for hyperkalemia).
Time Frame: First 7 days post-transplant
Measure: Count of Participants; unit: Participants
Groups:
- C1-Inhibitor (Berinert) (Human) (C1INH): 35 patients will receive C1 esterase inhibitor in addition to standard of care immunosuppressive therapy.
  C1 Esterase Inhibitor: C1 Esterase Inhibitor 50 units/kg IVPB administered on day of transplant, and another dose 24 hours post op. Total: 2 doses
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 34 | 35
Participants | 15 | 21

3. Primary Outcome: Number of Patients With Serum Creatinine Reduction Ratio of < 30% From 24 to 48 Hours Post-transplant.
Description: Number of patients in the C1INH and placebo groups with serum creatinine reduction of < 30% from 24 to 48 hours post-transplant.
Time Frame: First 7 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 35 | 35
Participants | 30 | 28

4. Primary Outcome: Number of Dialysis Sessions Per Patient in the First 7 Days Post Transplant.
Description: Mean quantity of dialysis sessions per patient in the first 7 days post transplant.
Time Frame: First 7 days post-transplant
Measure: Mean (Standard Deviation); unit: dialysis sessions
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 34 | 35
dialysis sessions | 0.97 (1.22) | 1.54 (1.54)

5. Secondary Outcome: Serum Creatinine
Description: Mean serum creatinine on day 90 in mg/dL
Time Frame: Up to 90 days post-transplant
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 35 | 35
mg/dL | 1.3 (0.317) | 1.7 (1.410)

6. Secondary Outcome: Creatinine Clearance
Description: Creatinine clearance calculated based on serum creatinine, milliliters per minute.
Time Frame: Up to 90 days post-transplant
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 35 | 34
ml/minute | 56.4 (15.558) | 51.2 (17.335)

7. Secondary Outcome: 24h Urine Output
Description: 24 hour urine output post-transplantation measured in milliliters
Time Frame: 24 hours post-transplant
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 35 | 35
milliliters | 873.5 (1257.0) | 607.8 (782.4)

8. Secondary Outcome: Mean Number of Patients on Dialysis
Description: Mean number of patients on dialysis at 15 to 30 days post-transplant
Time Frame: 15 to 30 days post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 35 | 35
Participants | 0 | 5

9. Secondary Outcome: Number of Patients With Delayed Graft Function (DGF) (Categorized by DGF Scale)
Description: DGF Scale:
  Grade 1 - immediate urine production and no need for dialysis with creatinine reduction ratio (CRR) between time 0 of transplantation and day 7 post-transplantation >70%
  Grade 2 - creatinine reduction ratio (CRR) between time 0 of transplantation and day 7 post-transplantation of >70% with need for dialysis
  Grade 3 - creatinine reduction ratio (CRR) between time 0 of transplantation and day 7 post-transplantation <70% with no need for dialysis
  Grade 4 - creatinine reduction ratio (CRR) between time 0 of transplantation and day 7 post-transplantation of <70% with need for dialysis.
Time Frame: First 7 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 34 | 35
Participants | 15 | 21

10. Other Pre Specified Outcome: Overall Incidence of Serious Adverse Events
Description: Overall incidence of serious adverse events in the C1INH and placebo groups, number of events.
Time Frame: Up to 9 months post-transplant
Measure: Number; unit: events
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 35 | 35
events | 11 | 16

11. Other Pre Specified Outcome: Patient Survival
Description: Patient survival at 90 days post-transplantation
Time Frame: Up to 90 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 35 | 35
Participants | 35 | 35

12. Other Pre Specified Outcome: Rate of Acute Cellular Rejection (ACR)
Description: Number of acute cellular and antibody mediated rejection episodes by day 90.
Time Frame: Up to 90 days post-transplant
Measure: Number; unit: episodes
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 35 | 35
episodes | 0 | 0

13. Other Pre Specified Outcome: Graft Survival
Description: Number of Participants with Graft Survival at 90 Days Post-Transplant
Time Frame: Day 90 Post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
Number analyzed (Participants) | 35 | 35
Participants | 34 | 34

ADVERSE EVENTS:
Time Frame: Adverse event data collected up to 9 months post transplant.
Arm/Group | C1-Inhibitor (Berinert) (Human) (C1INH) | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 10/35 | 10/35
Other Adverse Events (participants affected / at risk) | 28/35 | 26/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C1-Inhibitor (Berinert) (Human) (C1INH) (N=35) | Normal Saline (N=35)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Neutropenia/Fever (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Purulent Drainage from wound (Infections and infestations) | 1 (1) | 0 (0)
Acute Encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Sepsis from Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Endocrine disorders) | 1 (1) | 0 (0)
Flash pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
A fib, shortness of breath, chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Right leg DVT (Cardiac disorders) | 0 (0) | 1 (1)
Upper extermity/facial swelling, SVC syndrome (Cardiac disorders) | 0 (0) | 1 (1)
A flutter (Cardiac disorders) | 0 (0) | 1 (1)
Afib/ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Non ST segment elevation (Cardiac disorders) | 1 (1) | 0 (0)
Elevated creatinine/edema (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrectomy due to poor perfusion (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine Leak (Renal and urinary disorders) | 0 (0) | 1 (1)
Peri-renal transplant hematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Slurred speech/weakness/fatigue (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C1-Inhibitor (Berinert) (Human) (C1INH) (N=35) | Normal Saline (N=35)
Fatigue (General disorders) | 2 (2) | 5 (5) — Generalized fatigue described by the patient
Hyperglycemia (Endocrine disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (7) | 7 (7)
Hypertension (Cardiac disorders) | 1 (1) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (7)
Edema (Cardiac disorders) | 7 (7) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Hypotension (Cardiac disorders) | 1 (1) | 2 (2)
Shortness of Breath (Cardiac disorders) | 1 (1) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitations of this study include the small sample size and single-center performance. However, the patient population was balanced between the two groups and donor organ characteristics, including implantation biopsies, were similar.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT02134314/Prot_SAP_000.pdf